CLINICAL TRIAL: NCT00633737
Title: The Effects of Stress Reduction on Surgical Wound Healing: A Randomised Controlled Trial
Brief Title: The Effects of Stress Reduction on Surgical Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Wound healing study
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Wound Healing; Stress; Surgery
Keywords: Psychology; Laparoscopy; Cholecystectomy; Psychoneuroimmunology; Wound healing; Preparation for surgery; Stress reduction; Stress; Relaxation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stress reduction intervention
  Interventions: Behavioral: Stress reduction intervention
- 2 (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Stress reduction intervention — In addition to standard care, patients in the intervention group will receive a one-hour individually delivered programme administered once by a psychologist at least 3 days prior to surgery. This session aims to reduce stress and involves teaching relaxation and guided imagery exercises. Patients are provided a CD (or audiotape)of the relaxation instructions to take home and practice once a day.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate whether a stress reduction intervention prior to surgery can improve wound healing and recovery.The investigators hypothesise that patients who receive a psychological stress reduction intervention prior to surgery will report lower stress and higher perceived control, have lower stress hormones, better wound healing and better self-reported recovery than patients who receive standard care alone.

DETAILED DESCRIPTION:
In previous prospective research, psychological stress has been shown to slow the healing of small superficial wounds and impair surgical healing. We will investigate whether a psychological intervention to reduce stress can improve surgical healing.

Ninety patients undergoing elective laparoscopic cholecystectomy will be randomised to receive either standard care or a brief pre-surgical psychological intervention plus standard care. Patients will complete a pre-surgical questionnaire to assess stress, anxiety, depression, illness perceptions and current health, at least 3 days prior to surgery. Then the intervention will be delivered. A second questionnaire on the morning of surgery will reassess stress, anxiety and illness perceptions to see whether the intervention has reduced stress and increased control perceptions. Plasma catecholamines and salivary cortisol will be tested to assess the effectiveness of the intervention in reducing stress-related hormones and to investigate their role in wound healing. During surgery 2 small expanded polytetrafluroethylene tubes will be inserted in the wound, which will be removed after 7 days. Wound healing will be assessed by hydroxyproline and total protein deposition in the tubes, as well as by the presence of wound infection. Patients' post-surgical recovery, including pain and fatigue, will also be assessed. If this brief psychological intervention can improve wound healing and aid recovery, it would provide a simple strategy to improve outcomes in surgery.

ELIGIBILITY:
Inclusion Criteria:

* planned elective laparoscopic cholecystectomy at Manukau Surgical Centre
* able to understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
expanded polytetrafluoroethylene (ePTFE) tubes assessed for hydroxyproline deposited per unit length of the tube as well as total protein | 7 days following surgery

SECONDARY OUTCOMES:
Plasma catecholamines | morning of surgery, day after surgery, 7 days after surgery
Salivary cortisol | on morning before surgery (one sample). on day after surgery: samples immediately after waking, after 15 minutes, after 30 minutes and after 60 minutes
wound infection | 7 days after surgery
self-rated recovery (including fatigue, pain) | 7 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Broadbent, PhD, Principal Investigator — The University of Auckland
Locations (1):
- The University of Auckland, Auckland, New Zealand

REFERENCES:
- [Result] Broadbent E, Kahokehr A, Booth RJ, Thomas J, Windsor JA, Buchanan CM, Wheeler BR, Sammour T, Hill AG. A brief relaxation intervention reduces stress and improves surgical wound healing response: a randomised trial. Brain Behav Immun. 2012 Feb;26(2):212-7. doi: 10.1016/j.bbi.2011.06.014. Epub 2011 Jun 28. PMID 21741471
- [Result] Kahokehr A, Broadbent E, Wheeler BR, Sammour T, Hill AG. The effect of perioperative psychological intervention on fatigue after laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2012 Jun;26(6):1730-6. doi: 10.1007/s00464-011-2101-7. Epub 2012 Jan 19. PMID 22258294